CLINICAL TRIAL: NCT05503277
Title: A RANDOMIZED CONTROLED TRAIL COMARING LARYNGEAL TUBE SUCTION DISPOSABLE AND I-gel IN PEDIATRIC PATIENT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, MOSTAFA.SOMRI, Associate Clinical Professor of Anesthesiology, Bnai Zion Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 0117-22-BNZ
Record Dates: First submitted 2022-08-14; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Seal Pressure
Keywords: Supraglottic devices; ltsd; i-gel; pediatric; seal pressure

STUDY DESIGN:
Intervention Model Description: observational
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superglottic airway device LTSD (Active Comparator): measuring seal pressure
  Interventions: Device: LTSD
- Superglottic airway device i-gel (Active Comparator): measuring seal pressure
  Interventions: Device: i-gel

INTERVENTIONS:
Device: LTSD — measuring seal pressure
  Arms: Superglottic airway device LTSD
Device: i-gel — measuring seal pressure
  Arms: Superglottic airway device i-gel

SUMMARY:
Introduction The Laryngeal Tube Suction Disposable LTS-D and the i-gel are a second generation supraglottic airway device SAD, the devices have a drain tube to allow access to the gastrointestinal.

The i-gel is a second generation SAD. Does not need an inflatable cuff because the thermoplastic elastomer provides the seal.

The study designs to compare the Oropharyngeal leak pressure (OLP) of LTS-D with the i-gel that allow the use of Pressure Control Ventilation.

Materials and methods Approval obtained from the institute Ethics Committee, No 0117-22-BNZ. Written parental consent will be obtained Hundred children (50 patients in each device of both sex, weighing 10-35 kg, with an ASA physical status I, scheduled for elective minor surgery Study design Devices are the pediatric LTS-D and the i-gel. The patients will fast for 6 h for solids and 2 h for clear fluids and will be unpremeditated, anesthesia will initiate following a standardized protocol.

Both devices will be inserted blindly by expert pediatric anesthesiologists. Leak pressure, will be determined by closing the expiratory valve of the anesthesia breathing system and a fixed gas flow of 3 l min-1. The airway pressure at which an equilibrium is reached will be noted (maximum 40 cm H2O).

Primary outcome: Leak pressure Secondary outcome: SGAD insertion time Fiberoptic view Maneuvers Complications. Statistical Analysis the primary outcome is the leak pressure. Previous pilot conducted in 15 children, the average standard deviation leak pressure found to be 31 cm H20. In order to obtain a statistically representative sample for a 95% CI with a margin error of 2% and a standard deviation of 2 cm H20, the sample sizes of 50 cases are needed for each device.

Continuous data presented as mean±SD. For the categorical variables frequencies and percentages will be calculated. SPSS version 20 for statistical analysis. P-values smaller than 0.05 considered statistically significant.

Categorical data will be analyzed with Pearson chi-square test Mann-Whitney U test will be performed to analyze non-normally distributed interval scale data and ordinal categorical data. Normally distributed data will be analyzed by t-tests.

DETAILED DESCRIPTION:
Introduction The Laryngeal Tube Suction Disposable LTS-D and the i-gel are a second generation supraglottic airway device (SGA). A device have a drain tube to allow access to the gastrointestinal tract.

The LTS-D has recently undergone considerable changes in its design based on clinical studies users' feedback. It is available in all sizes, from newborn to adult.

The ventilation section between the proximal and distal cuff is significant different to the previous LTS-D. The ramp is conically shaped and increases space approximately 25% in the hypopharynx.

The i-gel is a second generation SAD, disposable airway is a SAD made of a medical grade thermoplastic elastomer. Its unique design does not need an inflatable cuff because the thermoplastic elastomer provides the seal. The i-gel is gaining a reputation for its ease of insertion and for its use in many clinical situations.

For our knowledge there are no published studies comparing the performances of the improved LTS-D and the i-gel in pediatric patients .

The study design to compare the Oropharyngeal leak pressure (OLP) of LTS-D with the i-gel that allow the use of Pressure Control Ventilation (PCV).

Materials and methods The Anesthesiology Department at the Bnai Zion Medical Center, Haifa, Israel, obtain the approval from the Local Ethics Committee, No 0117-22-BNZ.

Written parental consent will be obtained the surgery day. Data of 100 patients (50 patients in each device group) will be prospectively obtained. Patients are children of both sex, weighing 10-35 kg, with an ASA physical status I, and scheduled for elective minor surgery.

Patients will be excluded if their ASA physical status is II or more. Devices The devices are the pediatric LTS-D and the i-gel.

Study design The patients will fast for 6 h for solids and 2 h for clear fluids. All patients will be unpremeditated according with the Departmental policy. After installation of routine monitoring equipment, anesthesia will initiat following a standardized protocol. The anesthesia will be induced in a special pediatric induction room during parental presence by inhalation of sevoflurane and oxygen.

The patients in a supine position with the head on soft pillow. After the induction we will proceed to perform cannulation of a peripheral vein, and the patients will received fentanyl 2-3 μg kg-1 and propofol 3 mg kg-1. Neuromuscular block be produced by rocuronium bromide 0.6 mg/ֶkg and confirmed using a peripheral nerve stimulator Innervator, (Fisher& Paykel Electronic Ltd, Auckland, New Zealand) with a skin surface electrodes placed over the ulnar nerve, to elicit a motor response from the addutor pollicis brevis muscle. Train-of-four stimulation be monitored and insertion of the SGA will accomplished when the third twitch disappeared.

Maintenance of anesthesia conducted with 2-3% sevoflurane in 33 % oxygen and 66 % nitrous oxide and IV Fentanyl.

Both devices will be inserted in the "sniffing" position with the blind insertion technique as suggested per manufacture instruction by either two pediatric anesthesiologists who had used the Laryngeal Mask Airway ( LMA) more than 500 times and the LTS-D and i-gel more than 50 times in pediatric patients. The devices will be lubricated with a sterile jelly (K-Y gel, Johnson and Johnson, USA) The total time to achieve an effective airway will be measured as the time from removing the facemask until a normal square - wave capnograph tracing was observed.

Maneuvers If insertion of the device will allow some ventilation but judged inadequate by the above-described criteria, further maneuvers will be undertaken to properly position the device. These adjustments include minor interventions (adjusting head or neck position, applying jaw lift or gently pushing or pulling the device side to side ) or major interventions (reinsertion of or changing device size).

The easy of insertion will be graded as very easy, easy, difficult, or impossible.

Only two attempts at insertion will be allowed and if the two attempts unsuccessful the trachea will be intubated.

After insertion the cuffs of the LTS-D device will be inflated according to the manufacturer instructions using the original colored cuff syringe. The intracuff pressure (ICP) checked using a pressure gauge (VBM - Medizitechnik Sulz, Germany).

If the pressure is more than 60 cm H2O air will be removed in both sizes in order to obtain an optimal volume at a recommended value of 60 cm H2O intracuff pressure.

The intracuff pressure controlled by using a pressure gauge (VBM- Medizitechnik Sulz, Germany) Leak pressure, OLP determined by closing the expiratory valve of the anesthesia breathing system and a fixed gas flow of 3 l min-1. The airway pressure at which an equilibrium was reached was noted (maximum allowed 40 cm H2O).

Vocals cord view The fiberoptic position of the airway device will be determined according the technique proposing by Brimacombe J and Berry A by passing a 2.8-mm fiberoptic scope (Storz Gmbh, Tuttingen, Germany) to a position1 cm proximal to the ventilation holes of the SGD. The Score: 1= vocal cords not seen; 2 = vocal cords and anterior epiglottis visible; 3 = vocal cords and posterior epiglottis visible; 4 = only vocal cords visible.

The gastric tube Fr. 10 will be inserted through the dedicate device channel and the stomach will be empty from air and fluids. After the gastric sonda be removed, in an

attempt to assessed possible gastric insufflation, abdominal circumference will be measured at level of the umbilicus before the establishment of the PCV. This measure will be considered a baseline. And will be measured again at the end the surgery before the administration Atropine and Neostigmine.

The initial Inspiratory Pressure in cm H2O will be 15 cm H2O with a ventilation rate of 15 per min and inspiratory to expiratory time ratio (Ti:Te) was set at 1:2 and Peep 2 cmH2O. After the initial PCV a inspiratory pressure was increased or decreased, 1cm H2O in order to obtain an end tidal CO2 of 38-40 mmHg.

The following data will be recorded every 5 min commencing from the establishment of PCV until the neuromuscular block was abolished: oxygen saturation, end-tidal carbon dioxide, inspired and expired tidal volumes (TV ins., TV exp.) respiratory rate, compliance, inspiratory peak, plateau pressure and Peep. Systolic and diastolic blood

pressure and heard rate was too recorded before the induction and every 5 minutes during the surgery.

At end of surgery the neuromuscular blockade will be assessed by using train-of-four stimulation and all patients received Atropine 0.02mg/Kg and Neostigmine 0.04 mg/Kg to reverse residual neuromuscular block.

The airway device will be removed after the patients awakened to the point when they could open their mouth to command (or spontaneously). Each device will be examined for the presence of blood and the mouth was inspected for dental or mucosal trauma.

Baseline systolic BP (SBP), heart rate (HR) and Sp O2 will be recorded before insertion and then 1 and 5 min after insertion.

Perioperative adverse events related to the investigational device will be documented and graded as follows: mild = gagging on insertion; moderate = minimal blood staining of the device, sore throat, hoarseness, difficulty swallowing, severe = hypoxia, regurgitation, gastric insufflation and gross blood staining of the device. A research assistant will interview patients and their parents after release from the Post Anesthetic Care Unit (PACU) and again 24 h postoperatively by phone communication to determine the incidence of postoperative events.

The type of surgery will be minor Urology, Orthopedic and General Surgery of short and median duration.

Outcomes Measures Primary outcome

1. Leak pressure, OLP determined by closing the expiratory valve of the anesthesia breathing system and a fixed gas flow of 3 l min-1. The airway pressure at which an equilibrium was reached was noted (maximum allowed 40 cm H2O). (12)

   Secondary outcome SGAD insertion time The time taken from insertion of the SAD between the patient lips until the SAD is deemed to be correctly positioned by the participant by capnography and bilateral thorax auscultation of the lungs.
2. Fiberoptic view:

   Fiberoptic view rated according to the Fiber-Optic Scoring System proposed by Brimacombe et al. (13) in order to standardize the assessment of the SAD position (4 = only vocal cords seen; 3 = vocal cords plus posterior epiglottis seen; 2 = vocal cords plus anterior epiglottis seen; 1 = vocal cords not seen) evaluated by the investigator.
3. Maneuvers Maneuvers performed by the investigator on the SAD in order to visualized the vocal cord.

   Up-down Side to side ( left to right or right to left )
4. Complications

   Minor complications:

   Post Anesthesia Care Unit (PACU): blood staining on the device, soft tissue-trauma, sore throat, hoarseness, dysphonia difficulty in swallowing,

   Major complications:

   Aspiration, laryngospasm, oxygen desaturation (SpO2< 95), post extubation stridor
5. Subjective satisfaction of the participant about the performance of the devices

Following the study procedure, participants will be asked to complete a questionnaire independently and anonymously. They be asked to record the 'ease-of-use' of each technique, using a five-point Likert Scale (14) (''the tracheal tube with the fiberoptic was easily inserted into the trachea through which SAD''; 1 - strongly disagree, 2 - disagree, 3 - neither agree nor disagree, 4 - agree, 5 - strongly agree).

Data will be collected anonymously by a study investigator.

Successful in time insertion will be confirmed with the ability to achieve tidal volumes of at least 7 ml/kg with a square wave capnograph.

Statistical Analysis The primary outcome in this study was the leak pressure. Previous pilot conducted in 15 children, the average standard deviation leak pressure found to be 31 cm H20. In order to obtain a statistically representative sample for a 95% CI with a margin error of 2% and a standard deviation of 2 cm H20, the sample sizes of 50 cases are needed for each device/ Based on this calculation we included 50 patients in each group.

Continuous data are presented as mean±standard deviation. For the demographic continuous variables minimal and maximal values were calculated as well.

For the continuous variables "manometer values" and "leak pressure", 95% confidence intervals were calculated.

For the categorical variables frequencies and percentages were calculated. SPSS version 20 was used for statistical analysis. P-values smaller than 0.05 were considered statistically significant.

The abdominal circumference before and after the establishment of PCV will be analyzed by the Wilcoxon Signed Ranks test.

SPSS 28 (SPSS Inc., Chicago, IL) was used for statistical analysis and a P-value < 0.05 was considered statistically significant. Categorical data will be analyzed with Pearson chi-square test or with Fisher exact test, in case the expected values be smaller than 5. Mann-Whitney U test will be performed to analyze non-normally distributed interval scale data and ordinal categorical data. Normally distributed data will be analyzed by t-tests. Ordinal and categorical data be presented as number and percentage. Continuous normally distributed data be presented as mean± standard deviation (sd). Continuous non-normally distributed data are presented as mean±sd, median, range and [min, max]. The abdominal circumference before and after the establishment of PCV will be analyzed by the Wilcoxon Signed Ranks test

For the continuous variables "manometer values" and "leak pressure", 95% confidence intervals will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* ASA I
* ELECTIVE SURGRY

Exclusion Criteria:

* ASA II OR MORE
* At risk for aspiration
* Upper respiratory tract symptoms within former 10 days
* Congenital anatomical malformation
* A possible difficult airway by history or physical examination.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Seal pressure | 60 seconds
  Measuring seal pressure

SECONDARY OUTCOMES:
Device Insertion | 30 seconds
  Device insertion Time

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Somri, DR MD, Principal Investigator — Bnai Zion Medical Center

IPD SHARING:
Plan to Share IPD: No